CLINICAL TRIAL: NCT06516640
Title: Randomized Control Trial Evaluating the Impact of Continuous Glucose Monitoring Academy Education Curriculum Versus Standard Care on Glycemic Outcomes for Youth With Type 2 Diabetes
Brief Title: Type 2 Continuous Glucose Monitoring Academy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Barber, Rebecca, Nurse Scientist, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-24-00199; P50MD017344 (NIH)
Record Dates: First submitted 2024-06-11; First posted 2024-07-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Continuous Glucose Monitoring; Glycemic Control; Diabetes Education; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Receives standard of care, regular education in the clinic.
  Interventions: Behavioral: Standard Education
- Continuous Glucose Monitoring Academy (Experimental): Receive an interactive workbook with problem-based learning scenarios and video links about Continuous Glucose Monitoring and glucose management strategies (CGM Academy Program). Participate in four in-depth online group sessions with diabetes care and education specialists complete questionnaires three times: at the time of study enrollment, week 4 and 6 months.
  Interventions: Behavioral: Continuous Glucose Monitoring Academy; Behavioral: Standard Education

INTERVENTIONS:
Behavioral: Continuous Glucose Monitoring Academy — Educational materials as well as online sessions with diabetes educators.
  Arms: Continuous Glucose Monitoring Academy
Behavioral: Standard Education — Standard of care receives general education about diabetes.
  Other Names: Standard of Care

SUMMARY:
The goal of this clinical trial is to evaluate the Impact of Continuous Glucose Monitoring Academy Education Curriculum Versus Standard Care on Glycemic Outcomes for Youth With Type 2 Diabetes (T2D):

* The first aim is to determine how feasible it is to adapt the Continuous Glucose Monitoring Academy curriculum to teach youth with T2D glucose management strategies.
* The second aim is to evaluate the effects of the Continuous Glucose Monitoring Academy metrics.
* The third aim is to explore the relationships between these metrics with diabetes distress, diabetes family responsibilities, and process metrics.

Participants will join for a total of four weeks of education, followed by a six-month clinical review. They will have access to an online workbook and videos, and will participate in virtual sessions with a diabetes educator who will cover glucose management strategies in-depth. Participants will wear their preferred Continuous Glucose Monitoring system (Dexcom or FreeStyle Libre) provided via insurance and inserted at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Current age of 8-21 years;
2. T2D diagnosis;
3. Able to speak, read, and write English or Spanish

Exclusion Criteria:

a. Known history of medical adhesive allergies;

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in Time in Range (TIR) from baseline to 6 months | Baseline to 6 months
  Change in % glucose TIR (70-180 mg/dL)

SECONDARY OUTCOMES:
Mean change in Hemoglobin A1c (HbA1c) from baseline to 6 months | Baseline to 6 months
  Change in Hemoglobin A1c
Mean change in CGM metrics measured by CGM readings | Week 4 & 6 months
  % Glucose Time Below Range (<70mg/dL), % Glucose Time Above Range (>180mg/dL), % Glucose Variability (coefficient of variation, CV)
Change in perceived diabetes distress at baseline, week 4 & 6 months | Baseline, Week 4 & 6 months
  The Type 2 Diabetes Distress Assessment System (T2-DDAS) measures how much overall emotional distress is due to diabetes. Respondents are given statements about diabetes-related issues and indicate on a 5-point Likert scale (0 = not a problem, 1 = minor problem, 2 = moderate problem, 3 = somewhat serious problem, 4 = serious problem) the degree to which the statements are a problem. Increasing scores denote increased burden perceived.
Change in perceived diabetes family responsibility at baseline, week 4 & 6 months | Baseline, week 4 & 6 months
  The Diabetes Family Responsibility Questionnaire (DFRQ) is a 14-item validated survey assessing parental and child involvement in various diabetes management tasks. Youth and caregivers report on a 3-point scale (1=child, 2=equal, 3=parent) who is responsible for a given diabetes task. Higher scores indicate more parental involvement in diabetes management.
Average number of diabetes educator hours used per study participant at week 4 & 6 months. | Week 4 and 6 months
  Number of hours spent in diabetes education
Mean change in perceived benefits of Continuous Glucose (CGM) Monitor use | Week 4 & 6 months
  Name of questionnaire: Adolescent Benefits and Burdens of CGM Survey - BenCGM & BurCGM. Participants answer each question on a scale of Strong Disagree, Disagree, Neutral, Agree, Strongly Agree.
Mean change in perceived burden of Continuous Glucose Monitor (CGM) use | Week 4 & 6 months
  Name of questionnaire: Adolescent Benefits and Burdens of CGM Survey - BenCGM & BurCGM. Participants answer each question on a scale of Strong Disagree, Disagree, Neutral, Agree, Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Barber, PhD, RN, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No